CLINICAL TRIAL: NCT01796418
Title: Effect of Beraprost Sodium on Arterial Stiffness in Patients With Type 2 Diabetic Nephropathy (BESTinDN Study)
Brief Title: Beraprost Sodium and Arterial Stiffness in Patients With Type 2 Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Dong Ki Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BESTinDN-001
Record Dates: First submitted 2013-02-19; First posted 2013-02-21 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — beraprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beraprost sodium (Experimental): Beraprost sodium 0.02 mg capsule by mouth every 12 hours for 12 weeks
  Interventions: Drug: Beraprost sodium
- Placebo (Placebo Comparator): Placebo capsule by mouth every 12 hours for 12 weeks

INTERVENTIONS:
Drug: Beraprost sodium
  Other Names: Berasil
  Arms: Beraprost sodium

SUMMARY:
Diabetic nephropathy, the leading cause of end-stage renal disease in many countries, is characterized by high cardiovascular mortality and morbidity even in the early course of the disease. In addition, cardiovascular complication has been the most common cause of death in these patients. Thus, early detection and appropriate intervention for this highly common and critical complication is considered to play an important role in the management of the disease. In this regard, much interest has been focused on the early markers which can predict arterial diseases before the clinically apparent cardiovascular diseases. Recently, glowing evidence suggests that arterial stiffness as assessed by pulse wave velocity (PWV) may serve as a surrogate marker for future cardiovascular disease. In fact, increased PWV has been known to be independently associated with diabetic nephropathy in type 2 diabetes.

Beraprost sodium (BPS) is a stable orally active prostacyclin (PGI2) analogue that has a potent vasodilatory and anti-platelet effect. Also, BPS has been suggested to improve a micro-vascular circulation through a reduction of red blood cell deformability. In addition, recent studies have demonstrated that BPS improves endothelial function through an increase in endothelial nitric oxide synthesis and NO synthase gene transcription. These beneficial effects of BPS have been known to reduce PWV in patients prone to cardiovascular diseases such as elderly, hypertension, or a history of cerebral infarction. However, the effect of BPS on arterial stiffness in patients with diabetic nephropathy remains elusive. Our study will address the effect of BPS on arterial stiffness by PWV in patients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or more and 75 years or less
* Type 2 diabetes who is prescribed glucose-lowering agent or insulin
* Estimated glomerular filtration rate (GFR) by isotope dilution mass spectrometry (IDMS)- Modification of Diet in Renal Disease (MDRD) equation 30 ml/min/1.73 m2 or more
* verified 2 times or more of albuminuria 30 mg/g cr (or protein 300 mg/g cr)or more in a spot urine sample with interval of 1 week or more in recent 6 months
* Patients whose blood pressure is 140/90 mmHg or less and did not receive a prescription for additional antihypertensive medication in recent 3 months
* Patients who give written consent to this study by oneself

Exclusion Criteria:

* History of kidney transplantation
* current advanced congestive heart failure (NYHA class III or more)
* current uncontrolled arrhythmia
* current advanced liver cirrhosis (Child-Pugh class C)
* History of bleeding diathesis
* current active infection or uncontrolled inflammatory disorders
* History of cerebrovascular accident or myocardial infarction
* current use of anticoagulant
* current use of two or more antiplatelet agents
* patients with advanced malignancy (life expectancy less than 6 months)
* patients with uncontrolled diabetes (Hba1c more than 10%)
* patients with severe anemia (Hb less than 8.0 g/dL)
* female who are pregnant, trying to get pregnant or lactating
* Genetic diseases such as galactose intolerance, lactose deficiency or glucose-galactose malabsorption

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Brachial ankle pulse wave velocity (PWV) | 12 weeks
  The change of brachial ankle PWV at 12 weeks compared to baseline (0 week)

SECONDARY OUTCOMES:
Ankle brachial indices (ABI) | 12 weeks
  The change of ABI at 12 weeks compared to baseline (0 week)
Urine albumin creatinine ratio (UACR) | 12 weeks
  The change of UACR at 12 weeks compared to baseline (0 week)
IDMS MDRD estimated glomerular filtration rate (eGFR) | 12 weeks
  The change of IDMS MDRD eGFR at 12 weeks compared to baseline (0 week)
Lipid profiles | 12 weeks
  The change of total cholesterol, LDL-cholesterol, and triglyceride at 12 weeks compared to baseline (0 week)
Blood pressure | 12 weeks
  The change of systolic and diastolic blood pressure at 12 weeks compared to baseline (0 week)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Soo Lim, Prof, Study Chair — Department of Internal Medicine, Seoul National University Boramae Medical Center, Seoul, Korea; Dong Ki Kim, Prof, Principal Investigator — Department of Internal Medicine, Seoul National University Hospital, Seoul, Korea; Ki Young Na, Prof, Principal Investigator — Department of Internal Medicine, Seoul National University Bundang Hospital, Seongnam, Korea; Sung Gyun Kim, Prof, Principal Investigator — Hallym University Medical Center; Young-Ki Lee, Prof, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital
Locations (5):
- South Korea (5):
  - Hallym University Sacred Heart Hospital, Anyang
  - Seoul National University Bundang Hospital, Seongnam
  - Kangnam Sacred Heart Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Schiffrin EL, Lipman ML, Mann JF. Chronic kidney disease: effects on the cardiovascular system. Circulation. 2007 Jul 3;116(1):85-97. doi: 10.1161/CIRCULATIONAHA.106.678342. PMID 17606856
- [Background] Foley RN, Murray AM, Li S, Herzog CA, McBean AM, Eggers PW, Collins AJ. Chronic kidney disease and the risk for cardiovascular disease, renal replacement, and death in the United States Medicare population, 1998 to 1999. J Am Soc Nephrol. 2005 Feb;16(2):489-95. doi: 10.1681/ASN.2004030203. Epub 2004 Dec 8. PMID 15590763
- [Background] Melian EB, Goa KL. Beraprost: a review of its pharmacology and therapeutic efficacy in the treatment of peripheral arterial disease and pulmonary arterial hypertension. Drugs. 2002;62(1):107-33. doi: 10.2165/00003495-200262010-00005. PMID 11790158
- [Background] Sugawara A, Kudo M, Saito A, Matsuda K, Uruno A, Ito S. Novel effects of beraprost sodium on vasculatures. Int Angiol. 2010 Apr;29(2 Suppl):28-32. PMID 20357746
- [Background] Goya K, Otsuki M, Xu X, Kasayama S. Effects of the prostaglandin I2 analogue, beraprost sodium, on vascular cell adhesion molecule-1 expression in human vascular endothelial cells and circulating vascular cell adhesion molecule-1 level in patients with type 2 diabetes mellitus. Metabolism. 2003 Feb;52(2):192-8. doi: 10.1053/meta.2003.50025. PMID 12601631
- [Background] Nakayama T, Hironaga T, Ishima H, Maruyama T, Masubuchi Y, Kokubun S. The prostacyclin analogue beraprost sodium prevents development of arterial stiffness in elderly patients with cerebral infarction. Prostaglandins Leukot Essent Fatty Acids. 2004 Jun;70(6):491-4. doi: 10.1016/j.plefa.2003.10.004. PMID 15120711
- [Background] Nakayama T, Masubuchi Y, Kawauchi K, Masaki R, Hironaga T, Ishima H, Torigoe M, Shimabukuro H. Beneficial effect of beraprost sodium plus telmisartan in the prevention of arterial stiffness development in elderly patients with hypertension and cerebral infarction. Prostaglandins Leukot Essent Fatty Acids. 2007 Jun;76(6):309-14. doi: 10.1016/j.plefa.2007.05.004. Epub 2007 Jul 9. PMID 17616452
- [Background] Watanabe M, Nakashima H, Ito K, Miyake K, Saito T. Improvement of dyslipidemia in OLETF rats by the prostaglandin I(2) analog beraprost sodium. Prostaglandins Other Lipid Mediat. 2010 Sep;93(1-2):14-9. doi: 10.1016/j.prostaglandins.2010.04.003. Epub 2010 May 5. PMID 20450981
- [Background] Sato N, Kaneko M, Tamura M, Kurumatani H. The prostacyclin analog beraprost sodium ameliorates characteristics of metabolic syndrome in obese Zucker (fatty) rats. Diabetes. 2010 Apr;59(4):1092-100. doi: 10.2337/db09-1432. Epub 2010 Jan 12. PMID 20068136
- [Background] Rubin MF, Rosas SE, Chirinos JA, Townsend RR. Surrogate markers of cardiovascular disease in CKD: what's under the hood? Am J Kidney Dis. 2011 Mar;57(3):488-97. doi: 10.1053/j.ajkd.2010.08.030. Epub 2010 Dec 18. PMID 21168944
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915
- [Background] Noordzij M, Tripepi G, Dekker FW, Zoccali C, Tanck MW, Jager KJ. Sample size calculations: basic principles and common pitfalls. Nephrol Dial Transplant. 2010 May;25(5):1388-93. doi: 10.1093/ndt/gfp732. Epub 2010 Jan 12. PMID 20067907
- [Derived] Na KY, Kim DK, Kim SG, Lee YK, Lim CS. Effect of beraprost sodium on arterial stiffness in patients with type 2 diabetic nephropathy. Trials. 2013 Sep 2;14:275. doi: 10.1186/1745-6215-14-275. PMID 24066672